CLINICAL TRIAL: NCT05263180
Title: A First-in-human, Phase I Trial of EMB-09, a Bispecific Antibody Targeting PD-L1 and OX-40 in Patients With Advanced or Metastatic Solid Tumors
Brief Title: A Study of EMB-09 in Participants With Advanced or Metastatic Solid Tumors.
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai EpimAb Biotherapeutics Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EMB09X101
Record Dates: First submitted 2022-02-22; First posted 2022-03-02 (Actual); Last update posted 2023-10-18 (Actual); Status verified 2023-10

CONDITIONS: Advanced Solid Tumor
Keywords: Phase I; Bispecific antibody; OX40; PD-L1; EMB-09; Immuno-oncology; dose escalation; cohort expansion; advanced solid tumor

STUDY DESIGN:
Intervention Model Description: Single Group Assignment Dose escalation followed by Cohort Expansion Phase at the RP2D.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental: EMB-09 (Experimental): Participants enrolled at different time will receive EMB-09 once a week (IV) at different ascending dose levels.
  Interventions: Biological: EMB-09

INTERVENTIONS:
Biological: EMB-09 — EMB-09 is a FIT-Ig® bispecific antibody against PD-L1 and OX40.

SUMMARY:
This study is to evaluate the safety and tolerability of EMB-09 and to determine the maximum tolerated dose (MTD) and/or recommended Phase 2 dose (RP2D). Pharmacokinetics (PK), immunogenicity, and the anti-multiple myeloma activity of EMB-09 will also be assessed.

DETAILED DESCRIPTION:
This is a phase I, multi-center, open label, multiple dose, first in human study, designed to assess safety and tolerability, and to identify the maximum tolerated dose (MTD) and/or recommended Phase 2 dose for EMB-09 in patient with advanced or metastatic solid tumors. Pharmacokinetics,pharmacodynamics, immunogenicity and response will also be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide signed and dated informed consent prior to any study-related procedures and willing and able to comply with all study procedures.
* Phase I subjects:

  1. Patients with histologically or cytologically confirmed locally advanced/metastatic solid tumors including but not limited to melanoma, non-small cell lung cancer (NSCLC), triple negative breast cancer (TNBC), head and neck squamous cell carcinoma (HNSCC), nasopharyngeal cancer (NPC), hepatocellular carcinoma (HCC), gastric cancer (GC), endometrium cancer (EC), ovarian cancer (OC), renal cell carcinoma (RCC) and small cell lung cancer (SCLC), colorectal cancer (CRC).
  2. Patients who have failed (progressed on, or are intolerant of) standard therapies or no available standard treatment
  3. Measurable or evaluable disease per RECIST v1.1.
* Patients must provide archival tumor, or a fresh tumor biopsy will be required if archival tumor sample is not available. Archival tumor sample must be taken <2 years prior to screening, otherwise a fresh tumor biopsy at screening is required.
* ECOG performance status 0 or 1; life expectancy > 3 months.
* Adequate organ function to participate in the trial.
* Recovery from adverse events (AEs) related to prior anticancer therapy.
* Highly effective contraception

Exclusion Criteria:

* Patients who have active autoimmune disease or history of autoimmune disease
* History of severe irAE.
* History of severe allergic reactions
* Use of systemic corticosteroids.
* Symptomatic central nervous system metastases.
* Patients with cardiac dysfunction
* Uncontrolled diabetes mellitus with hemoglobin A1c > 8% (via medical history)
* Prior treatment with TNFRSF agonists including OX40, CD27, CD137 (4-1BB), CD357 (GITR), CD40.
* Anticancer therapy or radiation < 5 half-lives or 4 weeks (whichever is shorter) prior to study treatment;
* Current or history of idiopathic pulmonary fibrosis, interstitial lung disease, or organizing pneumonia.
* Concurrent malignancy < 5 years prior to entry.
* Patients with active infections.
* Major surgery < 4 weeks or minor surgery < 2 weeks prior to study treatment.
* Live virus vaccines < 30 days prior to screening
* Pregnant or breast-feeding females
* Any investigational agents or study drugs from a previous clinical study within 30 days of the first dose of study treatment.
* Any other serious underlying medical conditions
* Abuse of alcohol, cannabis-derived products, or other drugs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-07-25 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of adverse events as assessed by CTCAE V5.0 | Screening up to 30 days after the last dose.
  Incidence and severity of AE.
Incidence of serious adverse events. (SAE) | Screening up to 30 days after the last dose, or beyond 30 days if SAE is confirmed to be treatment related.
  Incidence of SAE.
Incidence of dose interruptions. | Screening up to 30 days after the las dose.
  Incidence of dose interruptions of EMB-09 during treatment as a measure of tolerability.
Dose intensity. | Screening up to 30 days after the last dose.
  Actual amount of drug taken by patients divided by the planned amount.
The incidence of DLTs during the first cycle of treatment. | First infusion to the end of cycle 1. (each cycle is 28 days)
  The dose limiting toxicities are based on drug related adverse events and are specifically defined in study protocol.

SECONDARY OUTCOMES:
Overall response rate | From the date of dosing until the date of first documented progression or date of death from any cause, whichever case first, expected average 6 months.
  Measured by RECIST 1.1.
Area under the serum concentration-time curve (AUC) of EMB-09 | Through treatment until EOT visit, expected average 6 months
  Blood samples for serum PK analysis will be obtained (AUC).
Maximum serum concentration (Cmax) of EMB-09 | Through treatment until EOT visit, expected average 6 months
  Blood samples for serum PK analysis will be obtained (Cmax)
Trough concentration (Ctrough) of EMB-09 | Through treatment until EOT visit, expected average 6 months
  Blood samples for serum PK analysis will be obtained (Ctrough)
Average concentration over a dosing interval (Css, avg)of EMB-09. | Through treatment until EOT visit, expected average 6 months
  Blood samples for serum PK analysis will be obtained (Css, avg).
Terminal half-life (T1/2) of EMB-09 | Through treatment until EOT visit, expected average 6 months
  Blood samples for serum PK analysis will be obtained (T1/2)
Systemic clearance (CL) of EMB-09 | Through treatment until EOT visit, expected average 6 months
  Blood samples for serum PK analysis will be obtained (CL).
Steady state volume of distribution (Vss) of EMB-09 | Through treatment until EOT visit, expected average 6 months
  Blood samples for serum PK analysis will be obtained (Vss).
Progression free survival (PFS) of EMB-09 as assessed by RECIST 1 | From the date of dosing until the date of first documented progression or date of death from any cause, whichever came first, expected average 6 months
  Preliminary anti-tumor activity of EMB-09 will be obtained. (DOR)
Incidence and titer of anti-drug antibodies stimulated by EMB-09 | Up to End of Treatment Follow Up Period (30 days after the last dose
  Antibodies to EMB-09 will be assessed to evaluate potential immunogenicity.

CONTACTS AND LOCATIONS:
Locations (4):
- Australia (3):
  - Peninsula and South Eastern Haematology & Oncology Group, Frankston
  - GenesisCareNorthShore, Leonards Hill
  - Blacktown Hospital, Sydney
- FUSCC, Shanghai, China

IPD SHARING:
Plan to Share IPD: No